CLINICAL TRIAL: NCT02529020
Title: Acute Effects of Jaw Clenching Using a Customized Mouthguard on Anaerobic Ability and Ventilatory Flows
Brief Title: Jaw Clenching on Anaerobic Ability and Ventilatory Flows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Responsible Party: Principal Investigator, Jose Morales, PHD, University Ramon Llull
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: mou01
Record Dates: First submitted 2015-08-11; First posted 2015-08-19 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Mouth Breathing
Keywords: mouthguard; ventilation; anaerobic power; ergogenic effects
MeSH Terms: conditions — Mouth Breathing; Respiratory Aspiration | interventions — Mouth Protectors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mouthguard (Experimental): All subjects perform all tests wearing mouthguard.
  Interventions: Device: Mouthguard
- No mouthguard (Experimental): All subjects perform all tests without mouthguard
  Interventions: Device: No mouthguard

INTERVENTIONS:
Device: Mouthguard — Condition of wearing mouthguard
  Arms: Mouthguard
Device: No mouthguard — Condition without mouthguard
  Arms: No mouthguard

SUMMARY:
The latest findings on the ergogenic effects of a dentistry-design, bite-aligning mouthpiece require additional research to assess its impact on anaerobic ability and ventilatory parameters. This study was aimed at determining the ergogenic acute effects of wearing a custom-made mouthpiece on oral airflow dynamics, Wingate Test performance parameters.

DETAILED DESCRIPTION:
The objectives of this study are to investigate the acute effects of a customized, bite-aligning mouthpiece on the different parameters assessed during a Wingate Test, as compared to clenching the jaw without a mouthpiece, in a physically-active, male population. The study also investigate the influence of wearing a mouthpiece on non-forced and forced airflow dynamics, as compared to open mouth and a jaw clenching without mouthpiece. Mouthpieces are made using a new scanning method that simplified the fitting process and lowered its cost.

A nonrandomized study was designed to compare the effect of the occlusion condition on the anaerobic power and airflow dynamics. Conditions of wearing or not wearing mouthguard (MOUTHG and NO-MOUTHG, respectively) are randomly distributed in all tests. Each subject participate in three sessions. The first session is used to obtain informed consent assess anthropometric measurements and to scan the subject's mouth structure. In the second session, subjects are familiarized with the test protocols via a learning session that included demonstration of Wingate Test and the airflow dynamics measurements. Subjects also perform the airflow tests and the first Wingate Test trial. In the third session, subjects perform the second Wingate Test trial. Conditions are randomly distributed in all tests. Wingate Test trials were separated by three days and subjects were not allowed to perform intensive training workloads.

ELIGIBILITY:
Inclusion Criteria:

* Healthy physical active males

Exclusion Criteria:

* Acute or chronic injury that caused pain during testing procedures
* Temporomandibular joint disorders

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in performance in Wingate test | 3 trials spaced 48 hours (each trial 30 seconds)
  Anaerobic power and capacity are assessed using the Wingate test with and without mouthguard (MOUTHG and NO-MOUTHG, respectively). Subjects complete a 30-sec maximal effort on an ergometer at a resistance equivalent to 7.5% of their body mass. The ergometer is interfaced with a computer loaded with software (Wingate Software Version 1.11, Lode BV) that apply the appropriate load for each subject. As a warm-up procedure, subjects are instructed to begin pedaling for 5 minutes at 100 W and approximately 60 rpm. After a 5 second count down and without altering the mentioned parameters, subjects are asked to begin pedaling as fast as possible while receiving verbal encouragement throughout the test. Peak power (W) and mean power (W) are calculated and recorded in an online data acquisition system.
Changes in performance dynamics airflow measurements. | 3 trials spaced 3 minutes (each trial 30 seconds)
  Subjects are asked to breath at resting pace during 30-sec under three different conditions: open mouth without mouthguard, jaw clenching without mouthguard and jaw clenched with mouthguard (OMNM, JCNM and JCM, respectively). Subjects intercalate 30 second forced breathings under the same conditions. Rest time was 3 minutes after both measurements under each condition. Conditions are randomly distributed. Facemask and is connected to a Biopac MP100 system through the wide-range airflow transducer amplifier. Peak air flow is detected and mean air flow during the 30 second interval is calculated for all conditions in L•min-1.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Pujades, PHD, Study Chair — Vicedagà Facultat ciències de l'Esport Blanquerna

REFERENCES:
- [Background] Arent, S. M., McKenna, J.and Golem, D. L. (2010). Effects of a neuromuscular dentistry-designed mouthguard on muscular endurance and anaerobic power. Comparative Exercise Physiology, 7(02), 73-79.
- [Background] Bailey SP, Willauer TJ, Balilionis G, Wilson LE, Salley JT, Bailey EK, Strickland TL. Effects of an over-the-counter vented mouthguard on cardiorespiratory responses to exercise and physical agility. J Strength Cond Res. 2015 Mar;29(3):678-84. doi: 10.1519/JSC.0000000000000668. PMID 25264671
- [Background] Cetin C, Kececi AD, Erdogan A, Baydar ML. Influence of custom-made mouth guards on strength, speed and anaerobic performance of taekwondo athletes. Dent Traumatol. 2009 Jun;25(3):272-6. doi: 10.1111/j.1600-9657.2009.00780.x. PMID 19583574